CLINICAL TRIAL: NCT06964425
Title: Raman Spectroscopy in the Diagnosis of Extrahepatic Cholangiocarcinoma
Brief Title: Raman Spectroscopy in the Diagnosis of Extrahepatic Cholangiocarcinoma - a Pilot Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Olomouc (Other)
Collaborators: Palacky University (Other)
Responsible Party: Principal Investigator, Peter Slodicka, Doctor of Medicine, Clinical Doctor, Principal Investigator, University Hospital Olomouc
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UHO005
Record Dates: First submitted 2025-04-15; First posted 2025-05-09 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Cholangiocarcinoma, Extrahepatic; Cholangiocarcinoma of the Extrahepatic Bile Duct; Cholangiocarcinoma, Perihilar; Diagnosis; Raman Spectroscopy; Klatskin Tumor; Endoscopy; Biliary Stricture; Malignant Biliary Stricture
MeSH Terms: conditions — Cholangiocarcinoma; Klatskin Tumor; Disease | interventions — Cholangiopancreatography, Endoscopic Retrograde

STUDY DESIGN:
Intervention Model Description: 20 patients with known extrahepatic cholangiocarcinoma, over 18 years of age
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- patients with extrahepatic cholangiocarcinoma (Experimental): 20 patients with known cholangiocarcinoma indicated for endoscopic retrograde cholangiopancreatography over 18 years of age
  Interventions: Procedure: Endoscopic retrograde cholangiopancreatography (ERCP)

INTERVENTIONS:
Procedure: Endoscopic retrograde cholangiopancreatography (ERCP) — Insertion of a endoscopic fiber-optic Raman probe under fluoroscopic control during endoscopic retrograde cholangiopancreatography to measure Raman spectra of extrahepatic cholangiocarcinoma and healthy bile duct.

SUMMARY:
Diagnosis of extrahepatic cholangiocarcinoma is challenging because the yield of imaging and tissue sampling is limited. Raman spectroscopy is an optical method based on the analysis of scattered monochromatic light. Raman spectroscopy is able to provide a molecular 'fingerprint' of the tissue to determine its type. The aim of this pilot study was to develop a methodology for in vivo Raman spectroscopy in bile ducts to improve the current diagnostic capabilities of extrahepatic cholangiocarcinoma.

DETAILED DESCRIPTION:
During ERCP, a fibre Raman probe (Endoscopic Fiber-Optic Raman Probe Bundle Fiber, Uni-Export Instruments, USA) is introduced transpapillary into the known extrahepatic cholangiocarcinoma. The Raman probe is placed in an adequate position under fluoroscopy control. Raman spectroscopy measurements are performed (without fluoroscopy) 20 times for each patient (laser wavelength 785 nm), 10 times for extrahepatic cholangiocarcinoma and 10 times for healthy bile duct. The attained data are saved and analysed by a specialised biophysicist. All patients provided informed consent.

ELIGIBILITY:
Inclusion Criteria:

* person older than 18 years, who has known extrahepatic cholangiocarcinoma and is indicated for ERCP

Exclusion Criteria:

* disagreement with the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-02-04 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
The differences in Raman spectra of malignant biliary tissue compared to healthy biliary tissue | Perioperative/Periprocedural
  During single ERCP procedure, we take 20 measurements of the Raman spectra (10 from malignant biliary tissue and 10 from healthy biliary tissue) that each tissue emits after interaction with the laser light. We are interested in the specific difference in the spectra of each tissue, which will be shown as a two-dimensional curve. The differences in the spectra of each tissue will be reflected by a change in the shape of the curve.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Slodička, M.D., Principal Investigator — University Hospital Olomouc
Locations (1):
- Peter Slodička, Olomouc, Olomoucký kraj, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Slodicka P, Falt P, Ranc V, Zoundjiekpon VD, Urban O. Raman spectroscopy in the diagnosis of malignant biliary stricture: A feasibility study. Hepatobiliary Pancreat Dis Int. 2025 Apr;24(2):211-216. doi: 10.1016/j.hbpd.2024.11.003. Epub 2024 Nov 16. No abstract available. PMID 39603958